CLINICAL TRIAL: NCT00676208
Title: Improving Medical Training for the Care of Chronic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SHP 08-141
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus
Keywords: Shared Medical Appointments; Diabetes; Education
MeSH Terms: conditions — Diabetes Mellitus | interventions — Shared Medical Appointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shared Medical Appointments (Experimental): Medical students participated in shared medical appointments for patients with diabetes for one month.
  Interventions: Behavioral: Shared Medical Appointments
- No shared medical appointments (No Intervention): Medical students in this arm did not participate in shared medical appointments.

INTERVENTIONS:
Behavioral: Shared Medical Appointments — Participated in shared appointments for patients as part of interprofessional team providing care for diabetes
  Arms: Shared Medical Appointments

SUMMARY:
While medical training has increasingly included chronic care management, quality care necessitates education approaches that go farther. In April 2005, the Louis Stokes Cleveland Veterans Affairs Medical Center (VAMC) implemented a weekly Diabetes Shared Medical Appointment (SMA). SMAs offer an important opportunity to improve chronic care and a unique setting for training physicians. In order to equip physicians with needed resources to manage chronic care, the ways in which SMA experiences are processed and integrated into learning about interdisciplinary approaches and expanding trainees' understanding of chronic care issues need to be examined.

DETAILED DESCRIPTION:
: Most physicians receive training in and about an acute care-oriented health care system that cannot adequately address the challenges of chronic care management. While medical training has increasingly included chronic care management, quality care necessitates education approaches that go farther. In April 2005, the Louis Stokes Cleveland VAMC implemented a weekly Diabetes Shared Medical Appointment (SMA). Results indicate that SMAs are sustained and, as such, SMAs offer an important opportunity to improve chronic care and a unique setting for training physicians. SMAs offer the potential to provide training in crucial skills that have to date remained less amendable to traditional educational practices. In order to equip physicians with resources to effectively and efficiently manage chronic care, the ways in which SMA experiences are processed and integrated into learning about interdisciplinary approaches and expanding trainees' understanding of chronic care issues need to be examined. Without addressing this gap, it is not possible to develop a comprehensive care model that links education and patient outcomes for chronic conditions, such as diabetes. Building on previous pilot work, we continued to address evaluating and validating instruments. The proposed pilot project included using a think-aloud protocol to evaluate and validate new items and scales assessing interdisciplinary team and chronic care/diabetes beliefs, and evaluating and adjusting direct observation coding tools for chronic condition care.

ELIGIBILITY:
Inclusion Criteria:

Medical Students:

Inclusion: All medical students participating in diabetes Shared Medical Appointment sessions or other training experiences during the course of the study.

Exclusion Criteria:

medical students who have participated in SMAs for patients with diabetes at the Cleveland VAMC in the past.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Aron, MD MS, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

REFERENCES:
- [Result] Watts SA, Gee J, O'Day ME, Schaub K, Lawrence R, Aron D, Kirsh S. Nurse practitioner-led multidisciplinary teams to improve chronic illness care: the unique strengths of nurse practitioners applied to shared medical appointments/group visits. J Am Acad Nurse Pract. 2009 Mar;21(3):167-72. doi: 10.1111/j.1745-7599.2008.00379.x. PMID 19302693

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Medical Students who are assigned to observe Shared Medical Appointments.
- Comparison: Medical students who do not experience Shared Medical Appointments during the study period April to August 2008.
Period: Overall Study
Arm/Group | Intervention | Comparison
Started | 14 | 19
Completed | 12 | 13
Not Completed | 2 | 6
Not completed — Lost to Follow-up | 0 | 2
Not completed — Incomplete data | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- SMA Participants: Medical Students who were assigned to observe Shared Medical Appointments (SMA).
- Comparison: Medical students who do not experience Shared Medical Appointments.
- Total: Total of all reporting groups
Arm/Group | SMA Participants | Comparison | Total
Number analyzed (Participants) | 14 | 19 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — Age of participants not relevant to study focus | NA — Age of participants not relevant to study focus | NA — Total not calculated because data are not available (NA) in one or more arms.
  Between 18 and 65 years | NA — Age of participants not relevant to study focus | NA — Age of participants not relevant to study focus | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | NA — Age of participants not relevant to study focus | NA — Age of participants not relevant to study focus | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex/Gender, Customized [Number; unit: participants]
  Not collected | NA — Gender of participants not relevant to study focus | NA — Gender of participants not relevant to study focus | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 19 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Confidence in Ability to Perform Teamwork
Description: A three item scale was used to assess confidence in ability to convey logic of recommendations to other providers, explain one's distinctive perspective, and be accountable to patients for a decision made by a colleague from another discipline. The responses for each item ranged from 'not at all confident' (0) to 'very confident' (4), with higher values indicating more confidence. The total scale ranged from 0 to 16 with higher being more confident. Difference scores were analyzed (post-pre) with positive and higher values indicating more favorable change.
Time Frame: Pre-intervention and Post-Intervention at 1 month
Measure: Mean (Standard Deviation); unit: units of a scale
Groups:
- SMA Participants: Medical students who are assigned to observe Shared Medical Appointments (SMA).
Arm/Group | SMA Participants | Comparison
Number analyzed (Participants) | 12 | 13
units of a scale | 1.40 (0.65) | -0.12 (0.6)
Statistical Analysis 1: Comparison: SMA Participants vs Comparison; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

2. Secondary Outcome: Change in Professionals' Attitudes About Diabetes
Description: The University of Michigan's Research and Training Center's Diabetes Attitude Scale was used. There are 33 items and the response format is a 5 point Likert Scale ranging from 'strongly disagree'(1) to 'strongly agree'(5). A higher score means more positive attitudes toward diabetes and its treatment (e.g., psychosocial impact of diabetes; value of tight glucose control).The total score is computed by summing individual items and ranges from 0 to 165. Post-pre total scores were used with positive and higher values indicating greater favorable change.
Time Frame: Pre-intervention and Post-intervention at 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- SMA Particiants: Medical students who were assigned to observe Shared Medical Appointments (SMA).
- Comparison: Medical students who do not experience Shared Medical Appointments (SMA).
Arm/Group | SMA Particiants | Comparison
Number analyzed (Participants) | 12 | 13
units on a scale | 0.88 (1.51) | -1.12 (2.85)
Statistical Analysis 1: Comparison: SMA Particiants vs Comparison; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | SMA Participants | Comparison
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/19
Other Adverse Events (participants affected / at risk) | 0/14 | 0/19

LIMITATIONS AND CAVEATS:
The small sample sizes and the reliance on one site for the data. This was a pilot study, both limitations were recognized from the outset and indeed seen as an advantage given the focus on trying to identify measures to include in a larger study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes